CLINICAL TRIAL: NCT03299959
Title: A Prospective Multicenter Open-label Randomized Controlled Trial of Agili-C™ vs. Surgical Standard of Care (SSOC) for the Treatment of Joint Surface Lesions of the Knee
Brief Title: Agili-C™ Implant Performance Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN0021
Record Dates: First submitted 2017-09-14; First posted 2017-10-03 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-11

CONDITIONS: Cartilage or Osteochondral Defects in the Knee; Up to Moderate Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Open-label Randomized Controlled Trial
Masking Description: Open-Label, adaptive design with interim analyses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Agili-C (Experimental)
  Interventions: Device: Agili-C implant
- Surgical Standard of Care (SSOC) (Active Comparator)
  Interventions: Procedure: SSOC

INTERVENTIONS:
Device: Agili-C implant — Agili-C implant
  Arms: Agili-C
Procedure: SSOC — microfracture and/or debridement
  Arms: Surgical Standard of Care (SSOC)

SUMMARY:
The current study compares the efficacy and safety of the Agili-C implant to Surgical Standard of Care treatment in patients suffering from joint surface lesions of the knee. The patient population is heterogeneous, involving different kinds of joint surface lesions: focal cartilage lesions, osteochondral defects and mild to moderate osteoarthritis, including multiple defects.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, randomized, and controlled trial of Agili-C™ vs. SSOC for the repair of joint surface lesions.

Follow-up visits will be performed at 2 weeks and at 3, 6, 12, 18, 24, 36, 48 and 60 months post-procedure to evaluate the patient's knee condition and clinical health.

The following questionnaires: KOOS, IKDC Knee Examination Form 2000, IKDC Subjective Knee Evaluation , SF-12 Health Survey, Tegner Activity Score will be completed at baseline and at 6, 12, 18, 24, 36, 48 and 60 months.

Anterior-Posterior (A/P) and Lateral knee X-rays will be taken at 2 weeks and at 6, 12, 18 24, 36, 48 and 60 months post procedure. MRI according to specific protocol will be performed at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. 21 -75 years
2. Up to 3 treatable joint surface lesion(s), ICRS Grade III or above, on the femoral condyles and/or trochlea
3. Symptomatic total treatable area 1-7 cm2. Asymptomatic lesions will not be included in the calculation
4. Must be physically and mentally willing and able to comply with the post-operative rehabilitation protocol and scheduled clinical and radiographic visits
5. Signed and dated the IRB/Ethics Committee approved Informed Consent Form and HIPPA (if applicable)
6. Non-responsive to physical therapy for at least 3-4 weeks

Exclusion Criteria:

1. KOOS Pain Subscale score at baseline is less than 20 or more than 65 (scale: maximum pain =0, pain free =100)
2. Bony defect depth deeper than 8mm, according to baseline MRI/X-ray/arthroscopy
3. Articular cartilage lesions in the tibia or the patella, ICRS grades IVa or above
4. Osteoarthritis of the index knee graded 4 according to the Kellgren-Lawrence Grading
5. Significant instability of the index knee according to IKDC Knee Examination Form 2000, Grade C (abnormal) or D (severely abnormal)
6. Malalignment more than 8 degrees varus OR 8 degrees valgus according to standing X-ray
7. Lack of functional remaining meniscus, at least 5mm rim at the end of the procedure
8. Meniscal transplantation in the past 6 months
9. Any known tumor of the index knee
10. Any known history of intra-articular or osseous infection of the index knee
11. Any evidence of active infection anywhere in the body. Urinary Tract Infection (UTI) patients can be included following antibiotic treatment, and provided that two consecutive cultures are negative (taken within at least 2 weeks of each other)
12. Any known history of inflammatory arthropathy or crystal-deposition arthropathy
13. Any known systemic cartilage and/or bone disorder, such as but not limited to, osteoporosis, chondrodysplasia or osteogenesis imperfecta
14. Body Mass Index (BMI) > 35
15. Chemotherapy in the past 12 months
16. Any previous surgical cartilage treatment (such as: microfracture, ACI, OATS, etc.) in the index knee within the last 6 months
17. Any previous ligamentous repair or malalignment correction in the index knee within the last 6 months
18. History of allergic reaction or intolerance of materials containing calcium carbonate or hyaluronate
19. Patient who is pregnant or intends to become pregnant during the study
20. History of any significant systemic disease, such as but not limited to: HIV, hepatitis, HTLV, syphilis, and coagulopathies
21. Known substance or alcohol abuse
22. Participation in other clinical trials within 60 days prior to the study or concurrent with the study
23. Known insulin dependent diabetes mellitus
24. Unable to undergo either MRI or X-ray
25. Use of anticoagulation medication or antiaggregant medication; however up to 100 mg Acetylsalicylic acid (ASA) daily is allowed
26. Previous intra-articular steroid injection within the last 1 month
27. Prisoners
28. Uncontained lesion - Lack of vital bone wall, at least 2mm thick, completely surrounding the lesion - based on MRI/X-ray/arthroscopy
29. Inability to position the implant 2mm recessed relative to the articular surface - based on MRI/X-ray/arthroscopy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, MD, Principal Investigator — Istituto Clinico Humanitas, Via A. Manzoni 56, Rozzano, Milano, Italy
Locations (26):
- United States (11):
  - Horizon Clinical Research, San Diego, California
  - LSU Healthcare Network Orthopedic & Sports Medicine, New Orleans, Louisiana
  - Peninsula Orthopaedic Associates, Salisbury, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Missouri, Missouri Orthopaedic Institute, Columbia, Missouri
  - NYU Langone Orthopedic Hospital, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Arlington Orthopedic Associates, Arlington, Texas
  - OrthoVirginia, Richmond, Virginia
- AZ Monica, Antwerp, Belgium
- Hungary (2):
  - Uzsoki Utcai Kórház, Budapest
  - Kastélypark Klinika, Tata
- Israel (5):
  - Assaf Harofeh Medical Center, Be’er Ya‘aqov
  - "Carmel" Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Hasharon Hospital, Petach Tikva, Petah Tikva
  - Souraski Medical Center, Tel Aviv
- Italy (2):
  - Humanitas Gavazzeni, Bergamo
  - Istituto Clinico Humanitas, Rozzano
- Specialist Hospital. Louis Rydygier in Krakow, Krakow, Poland
- County Hospital Timis Othopedy and Trauma Clinic, Timișoara, Romania
- Serbia (3):
  - Atlas General hospital, Belgrade
  - Clinic for Orthopedic Surgery "Banjica", Belgrade
  - Clinical Center of Vojvodina, Novi Sad

REFERENCES:
- [Derived] Kon E, De Caro F, Dasa V, M Scopp J, Di Matteo B, Flanigan D, Shabshin N, Strickland S, Altschuler N. Female patients report comparable results to males after the implantation of an aragonite-based scaffold for the treatment of knee chondral and osteochondral defects: a gender-based analysis of a RCT at 4 years' follow-up. J Orthop Traumatol. 2025 Mar 13;26(1):17. doi: 10.1186/s10195-025-00829-y. PMID 40080289
- [Derived] Altschuler N, Zaslav KR, Di Matteo B, Sherman SL, Gomoll AH, Hacker SA, Verdonk P, Dulic O, Patrascu JM, Levy AS, Robinson D, Kon E. Aragonite-Based Scaffold Versus Microfracture and Debridement for the Treatment of Knee Chondral and Osteochondral Lesions: Results of a Multicenter Randomized Controlled Trial. Am J Sports Med. 2023 Mar;51(4):957-967. doi: 10.1177/03635465231151252. Epub 2023 Feb 13. PMID 36779614

RESULTS

PARTICIPANT FLOW:
Groups:
- Agili-C™: Participants randomized to the investigational arm that received the Agili-C™ implant following arthroscopy via a mini-arthrotomy or arthrotomy approach
- Surgical Standard of Care (SSOC): Participants randomized to the control arm received surgical standard of care (SSOC) that included two procedures, microfracture (MFX) and debridement (Deb).
Period: Overall Study
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Started | 167 | 84
Completed | 130 | 57
Not Completed | 37 | 27
Not completed — Lost to Follow-up | 7 | 9
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 13 | 9
Not completed — Changes in study team and government regulations | 1 | 1
Not completed — Participant underwent surgical intervention in the index knee | 15 | 8

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included randomized participants that received treatment with Agili-C™ or Surgical Standard of Care (SSOC).
Groups:
- Total: Total of all reporting groups
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC) | Total
Number analyzed (Participants) | 167 | 84 | 251
Age, Customized [Count of Participants; unit: Participants] — Number of participants categorized by age in years as either ≥50 or <50
  Participants
    Age Category: ≥50 | 40 | 34 | 74
    Age Category: <50 | 127 | 50 | 177
Age, Customized [Count of Participants; unit: Participants] — Number of participants were categorized by age group as one of the following:
  * 21 to <45 (Young adulthood)
  * 45 to <65 (Middle adulthood)
  * ≥65 (Elderly)
  Participants
    Age Group: 21 to <45 (Young adulthood) | 94 | 41 | 135
    Age Group: 45 to <65 (Middle adulthood) | 68 | 40 | 108
    Age Group: ≥65 (Elderly) | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 33 | 93
  Male | 107 | 51 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 164 | 82 | 246
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 159 | 81 | 240
  Race: Black | 6 | 2 | 8
  Race: Asian | 1 | 0 | 1
  Race: Native | 1 | 0 | 1
  Race: Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: Participants]
  United States | 33 | 18 | 51
  Israel | 24 | 15 | 39
  Belgium | 6 | 2 | 8
  Poland | 6 | 3 | 9
  Hungary | 2 | 1 | 3
  Romania | 21 | 10 | 31
  Italy | 17 | 9 | 26
  Serbia | 58 | 26 | 84
Body Mass Index (BMI) ≥30 [Count of Participants; unit: Participants] — Participants with body mass index (BMI) greater than or equal to 30 kg/m²(Yes/No).
  Participants
    Yes | 37 | 27 | 64
    No | 130 | 57 | 187

OUTCOME MEASURES:

1. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Score Change From Baseline to 60 Months
Description: Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Score consists of 9 items. A Likert scale is used with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Scores are transformed to a 0 to 100 scale, with 0 representing a worse outcome and 100 representing a better outcome.
  The change from baseline score is reported as the mean of posterior distribution with 95% credible interval using the Bayesian model.
Time Frame: Baseline, 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline for the specified time frame.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 146 | 71
score on a scale | 37.71 [34.47 to 40.93] | 18.68 [13.89 to 23.43]

2. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QOL) Score Change From Baseline to 60 Months
Description: Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QOL) Score consists of 4 items. A Likert scale is used with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Scores are transformed to a 0 to 100 scale, with 0 representing a worse outcome and 100 representing a better outcome.
  The change from baseline score is reported as the mean of posterior distribution with 95% credible interval using the Bayesian model.
Time Frame: Baseline, 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 146 | 71
score on a scale | 45.22 [40.49 to 49.93] | 22.29 [15.53 to 29.15]

3. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Function in Daily Living (ADL) Score Change From Baseline to 60 Months
Description: Knee Injury and Osteoarthritis Outcome Score (KOOS) Function in Daily Living (ADL) Score consists of 17 items. A Likert scale is used with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Scores are transformed to a 0 to 100 scale, with 0 representing a worse outcome and 100 representing a better outcome.
  The change from baseline score is reported as the mean of posterior distribution with 95% credible interval using the Bayesian model.
Time Frame: Baseline, 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 146 | 71
score on a scale | 33.03 [29.84 to 36.18] | 16.45 [11.84 to 21.12]

4. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Symptoms Score Change From Baseline to 60 Months
Description: Knee Injury and Osteoarthritis Outcome Score (KOOS) Symptoms Score consists of 7 items. A Likert scale is used with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Scores are transformed to a 0 to 100 scale, with 0 representing a worse outcome and 100 representing a better outcome.
  The change from baseline score is reported as the mean of posterior distribution with 95% credible interval using the Bayesian model.
Time Frame: Baseline, 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 146 | 71
score on a scale | 30.52 [27.00 to 34.02] | 15.52 [10.38 to 20.72]

5. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Sports Score Change From Baseline to 60 Months
Description: Knee Injury and Osteoarthritis Outcome Score (KOOS) Sports Score consists of 5 items. A Likert scale is used with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Scores are transformed to a 0 to 100 scale, with 0 representing a worse outcome and 100 representing a better outcome.
  The change from baseline score is reported as the mean of posterior distribution with 95% credible interval using the Bayesian model.
Time Frame: Baseline, 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 146 | 71
score on a scale | 47.32 [42.46 to 52.18] | 25.11 [18.15 to 32.08]

6. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score Responder Rate Change From Baseline to 60 Months
Description: Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score consists of 5 subscales. A Likert scale is used with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Subscale scores are combined to produce the Overall Score that is transformed to a 0 to 100 scale, with 0 representing a worse outcome and 100 representing a better outcome. Responder rate was defined as the proportion of participants achieving ≥30-point improvement from baseline to 60 months in the KOOS Overall Score.
  The change from baseline data is reported as the mean of posterior distribution with 95% credible interval using the Bayesian model.
Time Frame: Baseline, 60 Months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 146 | 71
proportion of participants | 0.74 [0.67 to 0.81] | 0.34 [0.24 to 0.46]

7. Secondary Outcome: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months and 48 Months
Description: Change from Baseline to 36 Months and 48 months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, and 48 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates participants with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 150 | 73
score on a scale
  Change from Baseline to 36 Months | 41.4 (21.3) [-6.8 to 86.4] | 19.3 (19.2) [-7.8 to 55.7]
  Change from Baseline to 48 months: number analyzed (Participants) | 143 | 71
  Change from Baseline to 48 months | 41.9 (21.6) [0.0 to 86.4] | 17.3 (20.0) [-29.6 to 59.5]

8. Secondary Outcome: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Score Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in the International Knee Documentation Committee (IKDC) Subjective Evaluation score. The IKDC Score was developed to detect improvement or deterioration in symptoms, function, and sports activities due to knee impairment, including patients with meniscal injuries. The possible score ranges from 0 to 100, with a higher score indicating no limitation with daily or sporting activities and the absence of symptoms (i.e., a better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 150 | 73
score on a scale
  Change from Baseline to 36 Months | 41.1 (22.6) [-20.7 to 82.8] | 18.8 (20.6) [-11.5 to 71.3]
  Change from Baseline to 48 Months: number analyzed (Participants) | 144 | 71
  Change from Baseline to 48 Months | 41.6 (23.0) [-13.8 to 82.8] | 17.9 (21.3) [-16.1 to 69.0]
  Change from Baseline to 60 Months: number analyzed (Participants) | 146 | 71
  Change from Baseline to 60 Months | 41.0 (24.2) [-8.1 to 82.8] | 18.4 (21.9) [-13.8 to 70.1]

9. Secondary Outcome: Tegner Activity Scale Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Tegner activity scale. The Tegner activity scale was designed as a score of activity level to complement other functional scores for patients with ligamentous injuries. The Tegner activity scale is a numerical scale ranging from 0 to 10, with a higher score indicating higher levels of activity (i.e., a better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 150 | 73
score on a scale
  Change from Baseline to 36 Months | 2.3 (1.9) [-3 to 9] | 1.0 (1.5) [-1 to 8]
  Change from Baseline to 48 Months: number analyzed (Participants) | 144 | 71
  Change from Baseline to 48 Months | 2.2 (1.8) [-1 to 8] | 0.9 (1.6) [-2 to 8]
  Change from Baseline to 60 Months: number analyzed (Participants) | 146 | 71
  Change from Baseline to 60 Months | 2.1 (1.8) [-2 to 7] | 0.9 (1.7) [-2 to 8]

10. Secondary Outcome: Short Form Survey (SF-12) Physical Component Score Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in SF-12 Physical Component Score. The SF-12 Physical Component Score assesses health related quality of life. The score is on a scale ranging from 0 to 100, with a higher score indicating a better outcome.
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 150 | 73
score on a scale
  Change from Baseline to 36 Months | 15.4 (9.8) [-4.0 to 39.4] | 7.3 (10.9) [-18.4 to 40.3]
  Change from Baseline to 48 Months: number analyzed (Participants) | 144 | 71
  Change from Baseline to 48 Months | 15.5 (10.6) [-14.2 to 36.2] | 6.4 (10.9) [-14.8 to 38.7]
  Change from Baseline to 60 Months: number analyzed (Participants) | 146 | 71
  Change from Baseline to 60 Months | 15.2 (11.5) [-20.9 to 39.0] | 6.1 (11.0) [-16.3 to 42.2]

11. Secondary Outcome: Short Form Survey (SF-12) Mental Component Score Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in SF-12 Mental Component Score. The SF-12 Mental Component Score assesses mental health and well-being. The score is on a scale ranging from 0 to 100, with a higher score indicating a better outcome.
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 150 | 73
score on a scale
  Change from Baseline to 36 Months | 5.4 (12.8) [-23.2 to 36.4] | 1.7 (8.7) [-16.6 to 37.3]
  Change from Baseline to 48 Months: number analyzed (Participants) | 144 | 71
  Change from Baseline to 48 Months | 5.2 (12.9) [-23.5 to 38.1] | 1.7 (10.1) [-19.4 to 34.5]
  Change from Baseline to 60 Months: number analyzed (Participants) | 146 | 71
  Change from Baseline to 60 Months | 4.3 (13.7) [-27.7 to 36.4] | 1.4 (9.4) [-16.9 to 37.3]

12. Secondary Outcome: Chondral Lesions: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants with Chondral Lesions measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants that had chondral lesions with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 94 | 59
score on a scale
  Change from Baseline to 36 Months | 42.9 (21.3) [-6.8 to 86.4] | 19.8 (19.4) [-7.8 to 55.7]
  Change from Baseline to 48 Months: number analyzed (Participants) | 90 | 58
  Change from Baseline to 48 Months | 42.1 (23.1) [0.0 to 86.4] | 19.0 (19.3) [-1.5 to 59.5]
  Change from Baseline to 60 Months: number analyzed (Participants) | 91 | 58
  Change from Baseline to 60 Months | 41.3 (23.7) [-2.5 to 86.4] | 18.5 (20.1) [-0.6 to 64.1]

13. Secondary Outcome: Osteochondral Lesions: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants with Osteochondral Lesions measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants that had osteochondral lesions with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 56 | 14
score on a scale
  Change from Baseline to 36 Months | 39.0 (21.1) [-5.0 to 79.0] | 17.0 (18.8) [0.0 to 54.9]
  Change from Baseline to 48 Months: number analyzed (Participants) | 53 | 13
  Change from Baseline to 48 Months | 41.5 (19.0) [0.0 to 80.3] | 9.7 (21.7) [-29.6 to 55.4]
  Change from Baseline to 60 Months: number analyzed (Participants) | 55 | 13
  Change from Baseline to 60 Months | 36.6 (22.9) [0.0 to 80.5] | 10.0 (21.3) [-26.9 to 54.9]

14. Secondary Outcome: Single Lesion: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants with a Single Lesion measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants that had a single lesion with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 97 | 51
score on a scale
  Change from Baseline to 36 Months | 43.7 (19.6) [0.0 to 86.4] | 20.4 (19.5) [-1.0 to 55.7]
  Change from Baseline to 48 Months: number analyzed (Participants) | 93 | 49
  Change from Baseline to 48 Months | 43.8 (20.8) [0.0 to 86.4] | 18.5 (19.1) [-1.5 to 56.1]
  Change from Baseline to 60 Months: number analyzed (Participants) | 95 | 49
  Change from Baseline to 60 Months | 41.5 (22.5) [-2.5 to 86.4] | 17.8 (19.5) [0.0 to 56.3]

15. Secondary Outcome: Multiple Lesions: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants with Multiple Lesions measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants that had multiple lesions with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 53 | 22
score on a scale
  Change from Baseline to 36 Months | 37.3 (23.6) [-6.8 to 76.8] | 16.6 (18.7) [-7.8 to 53.7]
  Change from Baseline to 48 Months: number analyzed (Participants) | 50 | 22
  Change from Baseline to 48 Months | 38.4 (22.8) [0.0 to 78.0] | 14.7 (21.9) [-29.6 to 59.5]
  Change from Baseline to 60 Months: number analyzed (Participants) | 51 | 22
  Change from Baseline to 60 Months | 36.0 (24.9) [0.0 to 80.4] | 14.9 (22.6) [-26.9 to 64.1]

16. Secondary Outcome: Level of Osteoarthritis (Kellgren-Lawrence Grade 0-1): Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants based on their level of osteoarthritis measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
  Participants were categorized as without osteoarthritis based on Kellgren-Lawrence (K/L) grade of 0 to 1. K/L grading included Grade 0 (No evidence of osteoarthritis), Grade 1 (Doubtful), Grade 2 (Minimal), and Grade 3 (Moderate).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants with the specified level of osteoarthritis with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 83 | 25
score on a scale
  Change from Baseline to 36 Months | 42.5 (20.6) [0.0 to 86.4] | 20.4 (16.4) [-1.0 to 53.5]
  Change from Baseline to 48 Months: number analyzed (Participants) | 77 | 24
  Change from Baseline to 48 Months | 43.1 (21.7) [0.0 to 86.4] | 17.2 (15.7) [-1.5 to 43.2]
  Change from Baseline to 60 Months: number analyzed (Participants) | 79 | 24
  Change from Baseline to 60 Months | 39.4 (23.9) [0.0 to 86.4] | 14.3 (15.3) [0.0 to 48.1]

17. Secondary Outcome: Level of Osteoarthritis (Kellgren-Lawrence Grade 2-3): Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants based on their level of osteoarthritis measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
  Participants categorized with osteoarthritis based on Kellgren-Lawrence (K/L) grade of 2 to 3. K/L grading included Grade 0 (No evidence of osteoarthritis), Grade 1 (Doubtful), Grade 2 (Minimal), or Grade 3 (Moderate).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 67 | 48
score on a scale
  Change from Baseline to 36 Months | 40.1 (22.2) [-6.8 to 79.5] | 18.7 (20.7) [-7.8 to 55.7]
  Change from Baseline to 48 Months: number analyzed (Participants) | 66 | 47
  Change from Baseline to 48 Months | 40.5 (21.5) [0.0 to 79.5] | 17.3 (22.0) [-29.6 to 59.5]
  Change from Baseline to 60 Months: number analyzed (Participants) | 67 | 47
  Change from Baseline to 60 Months | 39.8 (23.0) [-2.5 to 80.4] | 18.2 (22.6) [-26.9 to 64.1]

18. Secondary Outcome: Total Lesion Area ≤3cm²: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants with a lesion area ≤3cm² measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants with the specified lesion area size with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 60 | 36
score on a scale
  Change from Baseline to 36 Months | 38.3 (20.3) [0.0 to 86.4] | 21.5 (17.8) [0.0 to 55.7]
  Change from Baseline to 48 Months: number analyzed (Participants) | 58 | 35
  Change from Baseline to 48 Months | 38.4 (21.1) [0.0 to 86.4] | 20.7 (19.3) [0.0 to 56.1]
  Change from Baseline to 60 Months: number analyzed (Participants) | 58 | 35
  Change from Baseline to 60 Months | 36.2 (22.1) [0.0 to 86.4] | 18.9 (19.6) [0.0 to 56.3]

19. Secondary Outcome: Total Lesion Area >3cm²: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants with a lesion area >3cm² measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 90 | 37
score on a scale
  Change from Baseline to 36 Months | 43.5 (21.8) [-6.8 to 79.5] | 17.1 (20.5) [-7.8 to 54.9]
  Change from Baseline to 48 Months: number analyzed (Participants) | 85 | 36
  Change from Baseline to 48 Months | 44.3 (21.7) [0.0 to 79.8] | 14.0 (20.3) [-29.6 to 59.5]
  Change from Baseline to 60 Months: number analyzed (Participants) | 88 | 36
  Change from Baseline to 60 Months | 41.8 (24.2) [-2.5 to 81.7] | 15.0 (21.3) [-26.9 to 64.1]

20. Secondary Outcome: Without Previous Ligament Reconstruction: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants without previous ligament reconstruction was measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants without previous ligament reconstruction with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 52 | 35
score on a scale
  Change from Baseline to 36 Months | 37.0 (24.3) [-6.8 to 79.0] | 18.1 (19.7) [-7.8 to 54.9]
  Change from Baseline to 48 Months: number analyzed (Participants) | 50 | 33
  Change from Baseline to 48 Months | 38.8 (24.7) [0.0 to 80.3] | 12.3 (19.1) [-29.6 to 59.5]
  Change from Baseline to 60 Months: number analyzed (Participants) | 51 | 33
  Change from Baseline to 60 Months | 35.5 (26.4) [0.0 to 81.7] | 11.8 (19.9) [-26.9 to 64.1]

21. Secondary Outcome: With Previous Ligament Reconstruction: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants with previous ligament reconstruction was measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants with previous ligament reconstruction with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 12 | 7
score on a scale
  Change from Baseline to 36 Months | 34.7 (19.9) [0.0 to 58.3] | 25.8 (23.1) [0.0 to 53.5]
  Change from Baseline to 48 Months | 31.9 (21.5) [0.0 to 56.1] | 23.4 (23.3) [0.0 to 53.5]
  Change from Baseline to 60 Months | 31.9 (21.9) [0.0 to 53.9] | 25.7 (24.6) [0.0 to 53.8]

22. Secondary Outcome: With Intact Meniscus: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants categorized by a meniscus status of intact meniscus (i.e., without a concomitant meniscectomy) was measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants in the meniscus status specified with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 85 | 38
score on a scale
  Change from Baseline to 36 Months | 41.9 (19.5) [0.0 to 79.0] | 20.9 (18.1) [-1.0 to 55.7]
  Change from Baseline to 48 Months: number analyzed (Participants) | 78 | 37
  Change from Baseline to 48 Months | 42.0 (20.1) [0.0 to 80.3] | 19.0 (19.4) [-1.5 to 56.1]
  Change from Baseline to 60 Months: number analyzed (Participants) | 81 | 37
  Change from Baseline to 60 Months | 40.7 (21.4) [-2.5 to 80.5] | 18.3 (19.1) [0.0 to 56.3]

23. Secondary Outcome: With Previous Partial Meniscectomy: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants categorized by a meniscus status of previous partial meniscectomy (i.e., with a prior meniscectomy) was measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 21 | 21
score on a scale
  Change from Baseline to 36 Months | 38.4 (26.2) [-6.8 to 75.8] | 14.5 (19.9) [-7.8 to 53.7]
  Change from Baseline to 48 Months | 38.5 (25.5) [0.0 to 79.8] | 11.3 (20.1) [-29.6 to 59.5]
  Change from Baseline to 60 Months | 38.3 (26.2) [0.0 to 81.7] | 11.7 (21.9) [-26.9 to 64.1]

24. Secondary Outcome: With Concomitant Partial Meniscectomy: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants categorized by a meniscus status of concomitant partial meniscectomy (i.e., with a concomitant meniscectomy) was measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 44 | 14
score on a scale
  Change from Baseline to 36 Months | 42.0 (22.3) [0.0 to 86.4] | 21.9 (211.3) [-6.6 to 54.9]
  Change from Baseline to 48 Months: number analyzed (Participants) | 44 | 13
  Change from Baseline to 48 Months | 43.4 (22.4) [0.0 to 86.4] | 22.2 (20.6) [0.0 to 53.5]
  Change from Baseline to 60 Months: number analyzed (Participants) | 44 | 13
  Change from Baseline to 60 Months | 38.1 (26.1) [0.0 to 86.4] | 21.3 (21.4) [-0.6 to 53.8]

25. Secondary Outcome: Active Pre-injury: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants categorized as active prior to injury (based on Tegner score) was measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants categorized as active pre-injury based on Tegner score with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 118 | 52
score on a scale
  Change from Baseline to 36 Months | 39.6 (21.0) [-6.8 to 86.4] | 20.2 (19.1) [-6.6 to 54.9]
  Change from Baseline to 48 Months: number analyzed (Participants) | 114 | 50
  Change from Baseline to 48 Months | 40.4 (21.1) [0.0 to 86.4] | 17.4 (20.2) [-29.6 to 59.5]
  Change from Baseline to 60 Months: number analyzed (Participants) | 117 | 50
  Change from Baseline to 60 Months | 38.0 (22.3) [-2.5 to 86.4] | 17.5 (21.1) [-26.9 to 64.1]

26. Secondary Outcome: Non-Active Pre-injury: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 36 Months, 48 Months, and 60 Months
Description: Change from Baseline to 36 Months, 48 Months, and 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score for participants categorized as non-active prior to injury (based on Tegner score) was measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Time Frame: Baseline, 36 Months, 48 Months, and 60 Months
Population: Full Analysis Set (FAS) consisted of all randomized participants with treatment in the Agili-C™ arm and in the SSOC arm with a valid KOOS overall score at baseline and at least one valid KOOS overall score post-baseline. Number analyzed in each row indicates only participants categorized as non-active pre-injury based on Tegner score with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 32 | 21
score on a scale
  Change from Baseline to 36 Months | 48.4 (21.2) [0.0 to 79.5] | 17.1 (19.8) [-7.8 to 55.7]
  Change from Baseline to 48 Months: number analyzed (Participants) | 29 | 21
  Change from Baseline to 48 Months | 48.0 (22.9) [0.0 to 79.8] | 17.1 (19.8) [0.0 to 56.1]
  Change from Baseline to 60 Months: number analyzed (Participants) | 29 | 21
  Change from Baseline to 60 Months | 46.0 (27.2) [0.0 to 81.7] | 15.6 (19.0) [0.0 to 56.3]

27. Primary Outcome: Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Baseline to 60 Months
Description: Change from Baseline to 60 Months in Knee Injury and Osteoarthritis Outcome Score (KOOS) Overall Score measured by the five subscales of Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items). A Likert scale is used for all items with five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the subscale scores are combined to calculate the KOOS Overall Score. The Overall Score is transformed to 0 to 100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
  The change from baseline score is reported as the mean of posterior distribution with 95% credible interval using the Bayesian model.
Time Frame: Baseline, 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
Number analyzed (Participants) | 146 | 71
score on a scale | 38.75 [35.22 to 42.25] | 19.52 [14.40 to 24.72]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from surgery through the end of study, approximately 60 months
Arm/Group | Agili-C™ | Surgical Standard of Care (SSOC)
All-Cause Mortality (participants affected / at risk) | 1/167 | 0/84
Serious Adverse Events (participants affected / at risk) | 49/167 | 25/84
Other Adverse Events (participants affected / at risk) | 120/167 | 68/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Agili-C™ (N=167) | Surgical Standard of Care (SSOC) (N=84)
coronary artery disease (Cardiac disorders) | 0 | 1
myocardial infarction (Cardiac disorders) | 0 | 1
conductive deafness (Ear and labyrinth disorders) | 1 | 0
abdominal hernia (Gastrointestinal disorders) | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 1
haemorrhoids (Gastrointestinal disorders) | 1 | 0
inguinal hernia (Gastrointestinal disorders) | 0 | 2
asthenia (General disorders) | 1 | 0
cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
cholelithiasis (Hepatobiliary disorders) | 1 | 0
allergy to metals (Immune system disorders) | 1 | 0
covid-19 (Infections and infestations) | 4 | 1
covid-19 pneumonia (Infections and infestations) | 1 | 0
ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
contusion (Injury, poisoning and procedural complications) | 4 | 0
hand fracture (Injury, poisoning and procedural complications) | 1 | 0
injury (Injury, poisoning and procedural complications) | 1 | 0
limb injury (Injury, poisoning and procedural complications) | 0 | 1
meniscus injury (Injury, poisoning and procedural complications) | 3 | 1
nerve injury (Injury, poisoning and procedural complications) | 0 | 1
post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
tendon rupture (Injury, poisoning and procedural complications) | 2 | 1
traumatic arthropathy (Injury, poisoning and procedural complications) | 1 | 0
ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
choroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
sciatica (Nervous system disorders) | 2 | 0
foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
device breakage (Product Issues) | 1 | 0
nephrolithiasis (Renal and urinary disorders) | 1 | 0
menometrorrhagia (Reproductive system and breast disorders) | 0 | 1
vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ligament operation (Surgical and medical procedures) | 1 | 1
thrombophlebitis (Vascular disorders) | 1 | 0
Decreased range of motion compared to baseline (Musculoskeletal and connective tissue disorders) | 1 | 0
Deep Vein Thrombosis (DVT) and related complications (Vascular disorders) | 0 | 1
Increased transient or chronic pain in the operated joint, compared to baseline (Musculoskeletal and connective tissue disorders) | 6 | 10
Infection & related symptoms (Infections and infestations) | 1 | 0 — Infection (including septicemia or deep infections in the operated joint) and related symptoms, such as fever and/or pus
Progression of osteoarthritis compared to baseline (Musculoskeletal and connective tissue disorders) | 0 | 2 — Progression of osteoarthritis (degeneration of surrounding bone and cartilage or delamination) compared to baseline
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Agili-C™ (N=167) | Surgical Standard of Care (SSOC) (N=84)
atrioventricular block second degree (Cardiac disorders) | 0 | 1
arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
middle ear effusion (Ear and labyrinth disorders) | 0 | 1
hypothyroidism (Endocrine disorders) | 1 | 0
secondary hypogonadism (Endocrine disorders) | 1 | 0
blepharospasm (Eye disorders) | 0 | 1
cataract (Eye disorders) | 1 | 1
eye irritation (Eye disorders) | 1 | 0
eye pain (Eye disorders) | 1 | 0
eyelid ptosis (Eye disorders) | 0 | 1
retinal vein occlusion (Eye disorders) | 1 | 0
vision blurred (Eye disorders) | 1 | 0
abdominal pain upper (Gastrointestinal disorders) | 1 | 0
anal fissure (Gastrointestinal disorders) | 1 | 0
anal fistula (Gastrointestinal disorders) | 0 | 1
colitis (Gastrointestinal disorders) | 0 | 1
colitis ulcerative (Gastrointestinal disorders) | 1 | 0
constipation (Gastrointestinal disorders) | 1 | 0
crohn's disease (Gastrointestinal disorders) | 0 | 1
diarrhoea (Gastrointestinal disorders) | 1 | 0
gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
inguinal hernia (Gastrointestinal disorders) | 1 | 0
umbilical hernia (Gastrointestinal disorders) | 1 | 0
adverse drug reaction (General disorders) | 0 | 1
chest pain (General disorders) | 0 | 1
influenza like illness (General disorders) | 0 | 1
thermal burn (General disorders) | 1 | 0
cholelithiasis (Hepatobiliary disorders) | 0 | 1
drug hypersensitivity (Immune system disorders) | 3 | 1
covid-19 (Infections and infestations) | 4 | 3
coxsackie viral infection (Infections and infestations) | 0 | 1
diverticulitis (Infections and infestations) | 1 | 0
ear infection fungal (Infections and infestations) | 1 | 0
folliculitis (Infections and infestations) | 0 | 1
gastroenteritis (Infections and infestations) | 2 | 0
influenza (Infections and infestations) | 1 | 0
molluscum contagiosum (Infections and infestations) | 1 | 0
nasopharyngitis (Infections and infestations) | 1 | 1
oesophageal candidiasis (Infections and infestations) | 1 | 0
onychomycosis (Infections and infestations) | 1 | 0
orchitis (Infections and infestations) | 1 | 0
otitis media (Infections and infestations) | 1 | 1
pharyngitis streptococcal (Infections and infestations) | 1 | 2
pneumonia (Infections and infestations) | 1 | 1
sinusitis (Infections and infestations) | 1 | 0
stitch abscess (Infections and infestations) | 1 | 0
suspected covid-19 (Infections and infestations) | 0 | 1
tooth abscess (Infections and infestations) | 1 | 0
tooth infection (Infections and infestations) | 0 | 1
upper respiratory tract infection (Infections and infestations) | 1 | 1
urinary tract infection (Infections and infestations) | 1 | 0
viral infection (Infections and infestations) | 1 | 0
animal bite (Injury, poisoning and procedural complications) | 1 | 0
cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
chemical burns of eye (Injury, poisoning and procedural complications) | 0 | 1
contusion (Injury, poisoning and procedural complications) | 2 | 4
epicondylitis (Injury, poisoning and procedural complications) | 0 | 2
facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
fall (Injury, poisoning and procedural complications) | 0 | 1
hand fracture (Injury, poisoning and procedural complications) | 1 | 0
head injury (Injury, poisoning and procedural complications) | 2 | 0
iatrogenic injury (Injury, poisoning and procedural complications) | 1 | 0
iliotibial band syndrome (Injury, poisoning and procedural complications) | 2 | 1
inadequate osteointegration (Injury, poisoning and procedural complications) | 1 | 0
joint injury (Injury, poisoning and procedural complications) | 2 | 0
ligament sprain (Injury, poisoning and procedural complications) | 5 | 0
limb fracture (Injury, poisoning and procedural complications) | 1 | 0
limb injury (Injury, poisoning and procedural complications) | 1 | 0
muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
muscle strain (Injury, poisoning and procedural complications) | 2 | 1
neck injury (Injury, poisoning and procedural complications) | 1 | 0
post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 1
procedural pain (Injury, poisoning and procedural complications) | 1 | 0
repetitive strain injury (Injury, poisoning and procedural complications) | 1 | 0
rib fracture (Injury, poisoning and procedural complications) | 1 | 1
road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
sciatic nerve injury (Injury, poisoning and procedural complications) | 0 | 1
skin laceration (Injury, poisoning and procedural complications) | 0 | 1
tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
abnormal weight gain (Metabolism and nutrition disorders) | 0 | 1
dehydration (Metabolism and nutrition disorders) | 0 | 1
gout (Metabolism and nutrition disorders) | 1 | 0
hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
obesity (Metabolism and nutrition disorders) | 1 | 0
type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 12
back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0
chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
haemarthrosis (Musculoskeletal and connective tissue disorders) | 3 | 1
intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 3 | 0
plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 | 1
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
tendon disorder (Musculoskeletal and connective tissue disorders) | 4 | 0
tendonitis (Musculoskeletal and connective tissue disorders) | 3 | 2
tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
giant cell tumour of tendon sheath (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
burning sensation (Nervous system disorders) | 1 | 0
carpal tunnel syndrome (Nervous system disorders) | 0 | 1
cervical radiculopathy (Nervous system disorders) | 1 | 0
migraine without aura (Nervous system disorders) | 0 | 1
peroneal nerve palsy (Nervous system disorders) | 1 | 0
post-traumatic headache (Nervous system disorders) | 0 | 1
sciatica (Nervous system disorders) | 10 | 5
syncope (Nervous system disorders) | 1 | 0
thoracic outlet syndrome (Nervous system disorders) | 1 | 0
haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
anxiety (Psychiatric disorders) | 0 | 1
claustrophobia (Psychiatric disorders) | 0 | 1
depression (Psychiatric disorders) | 1 | 0
dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
menometrorrhagia (Reproductive system and breast disorders) | 1 | 0
menopausal symptoms (Reproductive system and breast disorders) | 1 | 0
pelvic pain (Reproductive system and breast disorders) | 1 | 0
penile discharge (Reproductive system and breast disorders) | 1 | 0
prostatism (Reproductive system and breast disorders) | 1 | 0
vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0
bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 0
psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
rash (Skin and subcutaneous tissue disorders) | 1 | 0
skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
lymphoedema (Vascular disorders) | 1 | 0
phlebitis (Vascular disorders) | 1 | 0
thrombosis (Vascular disorders) | 1 | 0
varicose vein (Vascular disorders) | 1 | 0
Decreased range of motion compared to baseline (Musculoskeletal and connective tissue disorders) | 1 | 1
Increased swelling (or effusion) in the operated joint, compared to baseline (Musculoskeletal and connective tissue disorders) | 10 | 3
Increased transient or chronic pain in the operated joint, compared to baseline (Musculoskeletal and connective tissue disorders) | 31 | 31
Joint locking (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle atrophy compared to baseline (Musculoskeletal and connective tissue disorders) | 2 | 0
Progression of osteoarthritis compared to baseline (Musculoskeletal and connective tissue disorders) | 0 | 2 — Progression of osteoarthritis (degeneration of surrounding bone and cartilage or delamination) compared to baseline
Vascular damage (Vascular disorders) | 0 | 1
Wound complications (wound dehiscence, hematoma, site drainage or superficial infection) (Skin and subcutaneous tissue disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is the sponsor can review results communications before public release and can prohibit communications about trial results for less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor may request amendments or object to the publication. If requested, the PI will use best efforts to accept the incorporation into the publication any such amendments.

DOCUMENTS (2):
  • Study Protocol (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT03299959/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03299959/SAP_002.pdf